CLINICAL TRIAL: NCT06695364
Title: Namık Kemal Üniversitesi, Tıp Fakültesi, Aile Hekimliği AD,
Brief Title: Opinions of NKU Faculty of Medicine Interns and Intern Doctors on Distance Medicine Education During the Covid-19 Pandemic Period
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Eda ÇELİK GÜZEL, associate professor, Namik Kemal University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NKMJ-04809
Record Dates: First submitted 2024-08-01; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Qualitative Research
MeSH Terms: interventions — Longitudinal Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anket (Other): Not all classes were included in the study
  Interventions: Other: survey study

INTERVENTIONS:
Other: survey study — Not all classes were included in the study

SUMMARY:
Objective: Throughout world history, people in the pandemic have not only been in danger of their physical health but also seriously affected their mental health. To prevent the spread of the virus during the COVID-19 pandemic, the Council of Higher Education of our country has closed schools and conducted education and training via online education. Therefore, the anxiety, uncertainty and closure of schools by the epidemic caused anxiety. The aim of our study; The effect of the Covid-19 pandemic on medical faculty student education is to evaluate the satisfaction of students from distance education applications.

Material and Methods: Our study is a cross-sectional descriptive type and was conducted on 321 students studying in the 4th, 5th and 6th grades of Tekirdag Namık Kemal University Faculty of Medicine in the 2021-2022 academic year. A survey including students' sociodemographic characteristics and Distance Education Perspective (UEBA) was applied to collect data. The data were evaluated with statistical analysis.

Results: Of the participating students, 85 were in 4th-grade, 157 were in 5th-grade, 79 were 6th-grade medical students. Answers to the question "If there was a second choice, would you choose the Faculty of Medicine?" 119 stated that they would choose the medical faculty again, 102 stated that they would not, and 100 stated that they were undecided. Answers to the question "What is your preferred education system option from today" 17 of the students preferred only the online education system, 127 only the face-to-face education system, and 177 preferred the system with online and face-to-face education have stated.

Conclusion: In terms of students' answers to the survey, it was seen that their level of perspective on distance education was undecided and it was determined that many factors affected distance education satisfaction. As a result, medical faculty students' anxiety increased during the pandemic period and they were less satisfied with the distance education system.

Keywords: Medicine, pandemic, online education

ELIGIBILITY:
Inclusion Criteria Voluntary students enrolled in the 4th, 5th, and 6th grades of Tekirdağ Namık Kemal University Faculty of Medicine (FM) during the 2021-2022 academic year and who agreed to participate in the survey were included in the study.

Exclusion Criteria Students who did not meet the inclusion criteria (those in the 1st, 2nd, or 3rd grades or students from another university or faculty) were excluded from the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 321 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Opinions of NKU Faculty of Medicine Interns and Intern Doctors on Distance Medicine Education during the Covid-19 Pandemic Period | 3 year
  In the Title field, specify the measurement that will be used questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Namık kemal Üniversitesi tıp fakültesi Aile hekimliği AD., Tekirdağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
There is no issue with sharing all the data on our part.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code